CLINICAL TRIAL: NCT00010400
Title: Pilot Study of Cyclophosphamide in Patients With Life-Threatening Systemic Lupus Erythematosus or Antiphospholipid Antibody Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: 199/15673; JHOC-J9717; JHOC-97022128
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Systemic Lupus Erythematosus; Antiphospholipid Antibody Syndrome
Keywords: antiphospholipid antibody syndrome; arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Antiphospholipid Syndrome; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Cyclophosphamide; Filgrastim

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: filgrastim

SUMMARY:
OBJECTIVES:

I. Determine the induction of durable remission in patients with life-threatening systemic lupus erythematosus or antiphospholipid antibody syndrome treated with cyclophosphamide.

II. Determine the toxicity of this drug in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive cyclophosphamide IV on days 1-4 and filgrastim (G-CSF) beginning on day 10 and continuing until blood counts recover.

Patients are followed monthly for 6 months, and then every 3 months thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of life-threatening systemic lupus erythematosus (SLE); must show at least 4 American College of Rheumatology criteria for SLE; must have severe organ damage in 1 or more organs; must have 1 or more of the following indications of ongoing disease activity: disease activity score (SLEDAI) at least 4, hospitalization for disease activity within 12 months, life-threatening disease not captured on SLEDAI

OR

Diagnosis of antiphospholipid antibody syndrome by the Hughes criteria; must show severity by ongoing symptoms or signs of hypercoagulability in spite of warfarin therapy

--Patient Characteristics--

Hepatic: Bilirubin no greater than 2.0 mg/dL; transaminases no greater than 2.0 times normal

Renal: Creatinine no greater than 3.0 mg/dL

Cardiovascular: Ejection fraction at least 45%

Pulmonary: FVC, FEV1, or DLCO at least 50% predicted

Other: Not preterminal or moribund; not pregnant or nursing; fertile patients must use effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 1997-04

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Brodsky, Study Chair — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland

REFERENCES:
- [Derived] Petri M, Brodsky RA, Jones RJ, Gladstone D, Fillius M, Magder LS. High-dose cyclophosphamide versus monthly intravenous cyclophosphamide for systemic lupus erythematosus: a prospective randomized trial. Arthritis Rheum. 2010 May;62(5):1487-93. doi: 10.1002/art.27371. PMID 20131296